CLINICAL TRIAL: NCT02974790
Title: Diagnostic Performance of Echocardiography Performed by Emergency Physicians After a Basic Training
Acronym: ECHOBEDSIDE
Status: Terminated | Type: Observational
Why Stopped: Not enough patient
Sponsor: University Hospital, Limoges (Other)
Collaborators: University Hospital, Tours (Other)
Responsible Party: Sponsor
Other Study IDs: I16035 (ECHOBEDSIDE)
Record Dates: First submitted 2016-11-23; First posted 2016-11-28 (Estimated); Last update posted 2018-03-29 (Actual); Status verified 2018-03

CONDITIONS: Circulatory Failure; Echocardiography
Keywords: echocardiography; training; emergency department; circulatory failure
MeSH Terms: conditions — Shock; Emergencies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Circulatory failure: Patients with a circulatory failure due to a sepsis or not
  Interventions: Procedure: Echocardiography

INTERVENTIONS:
Procedure: Echocardiography — Two-dimensional imaging echocardiography

SUMMARY:
After a basic training to echocardiography, emergency physicians will have to answer simple clinical questions about circulatory failure mechanisms. The objective of the study is to assess the agreement between these answers and those of the expert physician in patients admitted in the emergency department with a circulatory failure due to sepsis or not. Emergency physicians will volunteer to take part in a basic training on echocardiography. The training will include 4 hours of theory, 2 hours of interactive clinical cases and 6 hours of tutored practice at patients' bedside (10 to 15 examinations). The objective of the practice sessions will be to learn the technical grounds of transthoracic echocardiography (TTE), the different views and to identify the anatomical structures. The second part of the study will start after the training. Each eligible patient will be successively assessed by two investigators: one emergency physician recently trained and the expert physician. The echocardiography will be performed as soon as possible in the emergency department before or after the initiation of treatment without delaying it. The order of hemodynamic assessments will be random depending on the availability of the investigators; both assessments will however be performed within 30 minutes. Each investigator will independently read the echocardiography in real time at patients' bedside. They will then answer a limited list of standardized questions using two-choice answers or predefined choices. Finally investigators will choose a therapeutic proposition among a predefined list based on the answers. Only the results of the echocardiography performed by the expert physician will be used in patient management.

DETAILED DESCRIPTION:
After a basic training to echocardiography, emergency physicians will have to answer simple clinical questions about circulatory failure mechanisms. The objective of the study is to assess the agreement between these answers and those of the expert physician in patients admitted in the emergency department with a circulatory failure due to sepsis or not. Emergency physicians will volunteer to take part in a basic training on echocardiography. The training will include 4 hours of theory, 2 hours of interactive clinical cases and 6 hours of tutored practice at patients' bedside (10 to 15 examinations). The objective of the practice sessions will be to learn the technical grounds of transthoracic echocardiography (TTE), the different views and to identify the anatomical structures. The second part of the study will start after the training. Each eligible patient will be successively assessed by two investigators: one emergency physician recently trained and the expert physician. The echocardiography will be performed as soon as possible in the emergency department before or after the initiation of treatment without delaying it. The order of hemodynamic assessments will be random depending on the availability of the investigators; both assessments will however be performed within 30 minutes. Each investigator will independently read the echocardiography in real time at patients' bedside. They will then answer a limited list of standardized questions using two-choice answers or predefined choices. Finally investigators will choose a therapeutic proposition among a predefined list based on the answers. Only the results of the echocardiography performed by the expert physician will be used in patient management.

ELIGIBILITY:
Inclusion Criteria:

* patients > 18 years old
* patients admitted in the Emergency Department of Limoges University Hospital
* patients with circulatory failure defined as 1 or more of the following criteria :
* clinical signs of tissue hypoperfusion
* mottling
* Encephalopathy
* Oliguria < 0.5 ml/kg/h
* biological signs of hypoperfusion
* Lactate > 2 mmol/L
* AND/OR Low blood pressure defined as a sBP < 90 mmHg or mBP < 65 mmHG or decrease of sBP > 40 mmHg compared with usual blood pressure
* OR Patients with signs of sepsis recently defined as the following :
* Suspicion of clinical infection
* At least 2 of the 3 following items (i.e. SOFA > 2 points with 1 point/item) :
* Glasgow score < 13
* Respiratory rate > 22 cycle/min
* Systolic blood pressure < 100 mmHg

Exclusion Criteria:

* Pregnant patients
* Moribund patients or with limited care
* Patients under legal protection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Hemodynamic assessment will target patients with circulatory failure and / or sepsis in emergency unit
Sampling Method: Probability Sample
Enrollment: 89 (Actual)
Dates: Start 2017-01-02 (Actual); Primary Completion 2018-01-02 (Actual); Study Completion 2018-03-02 (Actual)

PRIMARY OUTCOMES:
Agreement between emergency physician and referee physician echocardiography | Day 1
  Agreement between the measurements performed using two-dimensional imaging echocardiography by an emergency physician and the referring physician according to the following data :
  * size of the left ventricle
  * systolic function of the left ventricle
  * size of the right ventricle
  * dysfunction of the right ventricle
  * size of the inferior vena cava pericardial effusion

SECONDARY OUTCOMES:
Agreement between emergency physicians and referring physician therapeutic propositions | Day 1
  Agreement between emergency physicians and referring physician therapeutic propositions according to the following choices:
  * vascular filling define as a water volume of at least 500 mL
  * vasopressor support
  * positive inotropic therapy
  * salt and water depletion

CONTACTS AND LOCATIONS:
Locations (1):
- Limoges University Hospital, Limoges, France

IPD SHARING:
Plan to Share IPD: No